CLINICAL TRIAL: NCT03998501
Title: Do Cognitive Behavioral Therapy Skills Classes Increase a Resiliency-related Brain Connectivity Pattern to Posttraumatic Stress Disorder?
Brief Title: fMRI to Examine the Effect of CBTm to Increase Resiliency for PTSD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: University of Regina (Other)
Responsible Party: Principal Investigator, Ji Hyun Ko, PhD, Assistant Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HS22895
Record Dates: First submitted 2019-06-24; First posted 2019-06-26 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: 20 participants will receive 5-week CBTm intervention. The other 20 participants will be waitlisted, but they will undergo the same assessment at the same time. Assessment including MRI will be done before and after 5-week intervention and 3 months after.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): 5-week CBTm
  Interventions: Behavioral: Cognitive Behavioral Therapy with Mindfulness Class
- Waitlisted (No Intervention): Waitlisted (will receive 5-week CBTm 3 months after).

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy with Mindfulness Class — The CBTm classes are five, 90-minute sessions focused on strategies to reduce symptoms of anxiety and depression.
  Arms: Active

SUMMARY:
A substantial proportion of public safety personnel (PSP) develop service-related posttraumatic stress disorder (PTSD). PTSD is associated with a range of negative outcomes and its exact underlying neurophysiological mechanism is still not well understood. Cognitive behavioral therapy (CBT) is commonly prescribed to treat PTSD, and recent studies suggest that it may be effective in preventing the condition. We have developed a 5-session class focused on teaching introductory CBT skills to prevent and manage psychological distress, and we are currently in the process of launching a clinical trial to demonstrate its effectiveness in preventing PTSD and related conditions in PSP. In the proposed adjunctive study to this trial, we will quantitate the brain connectivity signature that is specific to the PTSD-resilience, and examine whether the classes increase this resilience-related brain mechanism.

DETAILED DESCRIPTION:
Our ultimate research goal is to develop and validate a preventive strategy for PTSD. We aim to 1) demonstrate neurophysiological evidence (using fMRI) of preventive CBTm classes for PTSD, and 2) validate the utility of the proposed imaging-based biomarker for PTSD-related resiliency. Emerging evidence suggests that a program such as CBTm classes could promote resiliency to PTSD in healthy individuals at high risk for trauma exposure. Further, our preliminary brain imaging data analysis suggests that we can quantitate the brain connectivity pattern that may reflect resilience to PTSD. We thus hypothesize that CBTm will increase the PTSD resilience-related brain connectivity pattern expression.

In this novel pilot imaging study, we will recruit 40 PSP without PTSD or other mental disorder from 120 participants participating in our larger clinical trial. Twenty will be from each arm (CBTm and wait-list). The effect of CBTm on fMRI-based measures will be compared between arms.

ELIGIBILITY:
Inclusion Criteria:

* Must be enrolled in our on-going parallel study - "Cognitive Behaviour Therapy with Mindfulness Course for Building Workplace Resilience: A Pilot Randomized Controlled Trial"

Exclusion Criteria:

* if they have received psychological or medication treatment for a mental disorder in the past 6 months or if they score above the clinical cutoff on the following self-report symptom measures: Posttraumatic Checklist-5 (PCL-5) score >37; Patient Health Questionnaire-9 (PHQ-9) score (depression) >10, Generalized Anxiety Disorder-7 (GAD-7) score >7, and the presence of suicidal ideation in the past six months. Individuals falling below these cutoff scores will receive further diagnostic assessment by a supervised PhD graduate student in Clinical Psychology. Those meeting criteria for PTSD or other mental disorder in the past 12 months as assessed by the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) or the Mini International Neuropsychiatric Interview (MINI v.7.0.2) will also be excluded. Finally, we will exclude individuals with any contraindication to MRI (e.g., claustrophobia and metal implants).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
PTSD resilience-related brain connectivity pattern scores | 1 hour
  fMRI-based graph theory pattern that was highly expressed in trauma-exposed control compared to PTSD and normal control. This method has not been published yet. The higher score are considered to be a better outcome (more resilience). It is a z-scored to the normal control dataset.
Connor-Davidson Resilience Scale | 1 month
  measure of resilience
Posttraumatic Checklist-5 | 1 month
  Symptoms of PTSD

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No